CLINICAL TRIAL: NCT00046280
Title: Multicenter AIDS Cohort Study (MACS)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: MACS
Record Dates: First submitted 2002-09-24; First posted 2002-09-26 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood serum, plasma, and cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a comprehensive observational study of HIV infection in homosexual and bisexual men.

DETAILED DESCRIPTION:
The Multicenter AIDS Cohort Study (MACS) provides important information about the changing nature of HIV-mediated disease progression, the impact of antiretroviral treatment, the nature of HIV pathogenesis, and viral and host genetic factors. This study will also assess the long-term patterns of therapy use and risk-taking behaviors.

Patients will have study visits every 6 months. The visits will include interviews, specimen collection, and a physical examination.

ELIGIBILITY:
Inclusion Criteria:

* HIV negative, or
* HIV positive and no history or current use of highly active antiretroviral therapy (HAART), or
* HIV positive HAART recipient with documentation of HAART initiation, no AIDS diagnosis prior to HAART initiation, and a CD4 cell count and HIV-1 RNA measurement within 6 months prior to first HAART use.
* Sexual intercourse with men or at least 5 male or female partners in the 5 years prior to enrollment.

Exclusion Criteria:

* Injection drug use within 1 year of enrollment.
* Perinatally acquired HIV infection.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Homosexual and bisexual men with and without HIV infection
Sampling Method: Probability Sample
Enrollment: 7087 (Estimated)
Dates: Start 1984-04; Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Public Health Center, Los Angeles, California
  - CORE Health Center, Chicago, Illinois
  - Johns Hopkins School of Public Health, Baltimore, Maryland
  - University of Pittsburgh School of Public Health, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Williams CF, Klinzman D, Yamashita TE, Xiang J, Polgreen PM, Rinaldo C, Liu C, Phair J, Margolick JB, Zdunek D, Hess G, Stapleton JT. Persistent GB virus C infection and survival in HIV-infected men. N Engl J Med. 2004 Mar 4;350(10):981-90. doi: 10.1056/NEJMoa030107. PMID 14999110
- [Result] Kingsley LA, Zhou SY, Bacellar H, Rinaldo CR Jr, Chmiel J, Detels R, Saah A, VanRaden M, Ho M, Munoz A. Temporal trends in human immunodeficiency virus type 1 seroconversion 1984-1989. A report from the Multicenter AIDS Cohort Study (MACS). Am J Epidemiol. 1991 Aug 15;134(4):331-9. doi: 10.1093/oxfordjournals.aje.a116094. PMID 1877593
- [Result] Margolick JB, Munoz A, Donnenberg AD, Park LP, Galai N, Giorgi JV, O'Gorman MR, Ferbas J. Failure of T-cell homeostasis preceding AIDS in HIV-1 infection. The Multicenter AIDS Cohort Study. Nat Med. 1995 Jul;1(7):674-80. doi: 10.1038/nm0795-674. PMID 7585150
- [Result] Jacobson LP, Kirby AJ, Polk S, Phair JP, Besley DR, Saah AJ, Kingsley LA, Schrager LK. Changes in survival after acquired immunodeficiency syndrome (AIDS): 1984-1991. Am J Epidemiol. 1993 Dec 1;138(11):952-64. doi: 10.1093/oxfordjournals.aje.a116815. PMID 7903022
- [Result] Munoz A, Xu J. Models for the incubation of AIDS and variations according to age and period. Stat Med. 1996 Nov 15-30;15(21-22):2459-73. doi: 10.1002/(sici)1097-0258(19961130)15:223.0.co;2-q. PMID 8931213
- [Result] Enger C, Graham N, Peng Y, Chmiel JS, Kingsley LA, Detels R, Munoz A. Survival from early, intermediate, and late stages of HIV infection. JAMA. 1996 May 1;275(17):1329-34. PMID 8614118
- [Result] Munoz A, Sabin CA, Phillips AN. The incubation period of AIDS. AIDS. 1997;11 Suppl A:S69-76. No abstract available. PMID 9451969
- [Result] Mellors JW, Munoz A, Giorgi JV, Margolick JB, Tassoni CJ, Gupta P, Kingsley LA, Todd JA, Saah AJ, Detels R, Phair JP, Rinaldo CR Jr. Plasma viral load and CD4+ lymphocytes as prognostic markers of HIV-1 infection. Ann Intern Med. 1997 Jun 15;126(12):946-54. doi: 10.7326/0003-4819-126-12-199706150-00003. PMID 9182471
- [Result] Lyles RH, Munoz A, Yamashita TE, Bazmi H, Detels R, Rinaldo CR, Margolick JB, Phair JP, Mellors JW. Natural history of human immunodeficiency virus type 1 viremia after seroconversion and proximal to AIDS in a large cohort of homosexual men. Multicenter AIDS Cohort Study. J Infect Dis. 2000 Mar;181(3):872-80. doi: 10.1086/315339. PMID 10720507
- [Result] Detels R, Tarwater P, Phair JP, Margolick J, Riddler SA, Munoz A; Multicenter AIDS Cohort Study. Effectiveness of potent antiretroviral therapies on the incidence of opportunistic infections before and after AIDS diagnosis. AIDS. 2001 Feb 16;15(3):347-55. doi: 10.1097/00002030-200102160-00008. PMID 11273215
- [Result] Tarwater PM, Mellors J, Gore ME, Margolick JB, Phair J, Detels R, Munoz A. Methods to assess population effectiveness of therapies in human immunodeficiency virus incident and prevalent cohorts. Am J Epidemiol. 2001 Oct 1;154(7):675-81. doi: 10.1093/aje/154.7.675. PMID 11581102
- [Result] Detels R, Munoz A, McFarlane G, Kingsley LA, Margolick JB, Giorgi J, Schrager LK, Phair JP. Effectiveness of potent antiretroviral therapy on time to AIDS and death in men with known HIV infection duration. Multicenter AIDS Cohort Study Investigators. JAMA. 1998 Nov 4;280(17):1497-503. doi: 10.1001/jama.280.17.1497. PMID 9809730
- [Result] Yamashita TE, Phair JP, Munoz A, Margolick JB, Detels R, O'Brien SJ, Mellors JW, Wolinsky SM, Jacobson LP. Immunologic and virologic response to highly active antiretroviral therapy in the Multicenter AIDS Cohort Study. AIDS. 2001 Apr 13;15(6):735-46. doi: 10.1097/00002030-200104130-00009. PMID 11371688
- [Result] Tarwater PM, Margolick JB, Jin J, Phair JP, Detels R, Rinaldo C, Giorgi J, Munoz A. Increase and plateau of CD4 T-cell counts in the 3(1/2) years after initiation of potent antiretroviral therapy. J Acquir Immune Defic Syndr. 2001 Jun 1;27(2):168-75. doi: 10.1097/00126334-200106010-00012. PMID 11404539
- [Result] Kleeberger CA, Phair JP, Strathdee SA, Detels R, Kingsley L, Jacobson LP. Determinants of heterogeneous adherence to HIV-antiretroviral therapies in the Multicenter AIDS Cohort Study. J Acquir Immune Defic Syndr. 2001 Jan 1;26(1):82-92. doi: 10.1097/00126334-200101010-00012. PMID 11176272
- [Result] Sacktor N, Lyles RH, Skolasky R, Kleeberger C, Selnes OA, Miller EN, Becker JT, Cohen B, McArthur JC; Multicenter AIDS Cohort Study. HIV-associated neurologic disease incidence changes:: Multicenter AIDS Cohort Study, 1990-1998. Neurology. 2001 Jan 23;56(2):257-60. doi: 10.1212/wnl.56.2.257. PMID 11160967
- [Result] Jacobson LP, Li R, Phair J, Margolick JB, Rinaldo CR, Detels R, Munoz A. Evaluation of the effectiveness of highly active antiretroviral therapy in persons with human immunodeficiency virus using biomarker-based equivalence of disease progression. Am J Epidemiol. 2002 Apr 15;155(8):760-70. doi: 10.1093/aje/155.8.760. PMID 11943695
- [Result] Munoz A, Kirby AJ, He YD, Margolick JB, Visscher BR, Rinaldo CR, Kaslow RA, Phair JP. Long-term survivors with HIV-1 infection: incubation period and longitudinal patterns of CD4+ lymphocytes. J Acquir Immune Defic Syndr Hum Retrovirol. 1995 Apr 15;8(5):496-505. doi: 10.1097/00042560-199504120-00010. PMID 7697447
- [Result] Phair JP, Mellors JW, Detels R, Margolick JB, Munoz A. Virologic and immunologic values allowing safe deferral of antiretroviral therapy. AIDS. 2002 Dec 6;16(18):2455-9. doi: 10.1097/00002030-200212060-00011. PMID 12461420
- [Result] Anastos K, Gange SJ, Lau B, Weiser B, Detels R, Giorgi JV, Margolick JB, Cohen M, Phair J, Melnick S, Rinaldo CR, Kovacs A, Levine A, Landesman S, Young M, Munoz A, Greenblatt RM. Association of race and gender with HIV-1 RNA levels and immunologic progression. J Acquir Immune Defic Syndr. 2000 Jul 1;24(3):218-26. doi: 10.1097/00126334-200007010-00004. PMID 10969345
- [Result] Silverberg MJ, Smith MW, Chmiel JS, Detels R, Margolick JB, Rinaldo CR, O'Brien SJ, Munoz A. Fraction of cases of acquired immunodeficiency syndrome prevented by the interactions of identified restriction gene variants. Am J Epidemiol. 2004 Feb 1;159(3):232-41. doi: 10.1093/aje/kwh036. PMID 14742283
- [Result] Riddler SA, Smit E, Cole SR, Li R, Chmiel JS, Dobs A, Palella F, Visscher B, Evans R, Kingsley LA. Impact of HIV infection and HAART on serum lipids in men. JAMA. 2003 Jun 11;289(22):2978-82. doi: 10.1001/jama.289.22.2978. PMID 12799406
- [Result] Cole SR, Hernan MA, Robins JM, Anastos K, Chmiel J, Detels R, Ervin C, Feldman J, Greenblatt R, Kingsley L, Lai S, Young M, Cohen M, Munoz A. Effect of highly active antiretroviral therapy on time to acquired immunodeficiency syndrome or death using marginal structural models. Am J Epidemiol. 2003 Oct 1;158(7):687-94. doi: 10.1093/aje/kwg206. PMID 14507605
- [Result] Sacktor N, Skolasky RL, Tarwater PM, McArthur JC, Selnes OA, Becker J, Cohen B, Visscher B, Miller EN; Multicenter AIDS Cohort Study (MACS). Response to systemic HIV viral load suppression correlates with psychomotor speed performance. Neurology. 2003 Aug 26;61(4):567-9. doi: 10.1212/01.wnl.0000076477.71313.6e. PMID 12939443
- [Result] Farinpour R, Miller EN, Satz P, Selnes OA, Cohen BA, Becker JT, Skolasky RL Jr, Visscher BR. Psychosocial risk factors of HIV morbidity and mortality: findings from the Multicenter AIDS Cohort Study (MACS). J Clin Exp Neuropsychol. 2003 Aug;25(5):654-70. doi: 10.1076/jcen.25.5.654.14577. PMID 12815503
- [Result] Thio CL, Seaberg EC, Skolasky R Jr, Phair J, Visscher B, Munoz A, Thomas DL; Multicenter AIDS Cohort Study. HIV-1, hepatitis B virus, and risk of liver-related mortality in the Multicenter Cohort Study (MACS). Lancet. 2002 Dec 14;360(9349):1921-6. doi: 10.1016/s0140-6736(02)11913-1. PMID 12493258
- [Result] Seage GR 3rd, Losina E, Goldie SJ, Paltiel AD, Kimmel AD, Freedberg KA. The relationship of preventable opportunistic infections, HIV-1 RNA, and CD4 Cell counts to chronic mortality. J Acquir Immune Defic Syndr. 2002 Aug 1;30(4):421-8. doi: 10.1097/00042560-200208010-00008. PMID 12138349
- [Result] Tam HK, Zhang ZF, Jacobson LP, Margolick JB, Chmiel JS, Rinaldo C, Detels R. Effect of highly active antiretroviral therapy on survival among HIV-infected men with Kaposi sarcoma or non-Hodgkin lymphoma. Int J Cancer. 2002 Apr 20;98(6):916-22. doi: 10.1002/ijc.10274. PMID 11948473
- [Result] Tang J, Shelton B, Makhatadze NJ, Zhang Y, Schaen M, Louie LG, Goedert JJ, Seaberg EC, Margolick JB, Mellors J, Kaslow RA. Distribution of chemokine receptor CCR2 and CCR5 genotypes and their relative contribution to human immunodeficiency virus type 1 (HIV-1) seroconversion, early HIV-1 RNA concentration in plasma, and later disease progression. J Virol. 2002 Jan;76(2):662-72. doi: 10.1128/jvi.76.2.662-672.2002. PMID 11752157
- [Result] Skolasky RL, Phair J, Detels R, Riddler S, Margolick J, Jacobson LP. Thrush and fever as markers of immune competence in the era of highly active antiretroviral therapy. AIDS Res Hum Retroviruses. 2001 Sep 20;17(14):1311-6. doi: 10.1089/08892220152596551. PMID 11602040
- [Result] Sacktor N, Tarwater PM, Skolasky RL, McArthur JC, Selnes OA, Becker J, Cohen B, Miller EN; Multicenter for AIDS Cohort Study (MACS). CSF antiretroviral drug penetrance and the treatment of HIV-associated psychomotor slowing. Neurology. 2001 Aug 14;57(3):542-4. doi: 10.1212/wnl.57.3.542. PMID 11502933
- [Result] Lau B, Gange SJ, Phair JP, Riddler SA, Detels R, Margolick JB. Use of total lymphocyte count and hemoglobin concentration for monitoring progression of HIV infection. J Acquir Immune Defic Syndr. 2005 Aug 15;39(5):620-5. PMID 16044017
- [Result] Chu H, Gange SJ, Yamashita TE, Hoover DR, Chmiel JS, Margolick JB, Jacobson LP. Individual variation in CD4 cell count trajectory among human immunodeficiency virus-infected men and women on long-term highly active antiretroviral therapy: an application using a Bayesian random change-point model. Am J Epidemiol. 2005 Oct 15;162(8):787-97. doi: 10.1093/aje/kwi268. Epub 2005 Aug 31. PMID 16135508
- [Result] Li X, Margolick JB, Conover CS, Badri S, Riddler SA, Witt MD, Jacobson LP. Interruption and discontinuation of highly active antiretroviral therapy in the multicenter AIDS cohort study. J Acquir Immune Defic Syndr. 2005 Mar 1;38(3):320-8. PMID 15735452
- [Result] Schneider MF, Gange SJ, Williams CM, Anastos K, Greenblatt RM, Kingsley L, Detels R, Munoz A. Patterns of the hazard of death after AIDS through the evolution of antiretroviral therapy: 1984-2004. AIDS. 2005 Nov 18;19(17):2009-18. doi: 10.1097/01.aids.0000189864.90053.22. PMID 16260908
- [Result] Modi WS, Scott K, Goedert JJ, Vlahov D, Buchbinder S, Detels R, Donfield S, O'brien SJ, Winkler C. Haplotype analysis of the SDF-1 (CXCL12) gene in a longitudinal HIV-1/AIDS cohort study. Genes Immun. 2005 Dec;6(8):691-8. doi: 10.1038/sj.gene.6364258. PMID 16177829
- [Derived] Minhas AS, Post WS, Liu B, Doria De Vasconcellos H, Haberlen SA, Feinstein M, Stosor V, Budoff M, Chew KW, Magnani JW, Brown T, Lima JAC, Wu KC. Association of HIV Serostatus and Inflammation With Ascending Aortic Size. J Am Heart Assoc. 2022 Mar 15;11(6):e023997. doi: 10.1161/JAHA.121.023997. Epub 2022 Mar 5. PMID 35253450
- [Derived] Haley DF, Edmonds A, Ramirez C, French AL, Tien P, Thio CL, Witt MD, Seaberg EC, Plankey MW, Cohen MH, Adimora AA. Direct-Acting Antiviral Hepatitis C Treatment Cascade and Barriers to Treatment Initiation Among US Men and Women With and Without HIV. J Infect Dis. 2021 Jun 15;223(12):2136-2144. doi: 10.1093/infdis/jiaa686. PMID 33141170